CLINICAL TRIAL: NCT04752514
Title: Prevalence of Dynamic Instability Among Football Players in the UAE: A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, lecturer of physical therapy, Delta University for Science and Technology
Other Study IDs: dynamic instability
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Football Players

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the purpose of this study is to determine dynamic instability prevalence in United Arab Emirates football players.

ELIGIBILITY:
Inclusion Criteria:

* male
* 16-24 years .

Exclusion Criteria:

* previous injury in lower extremities

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 200 male football players aged from 16 to 24 years old were recruited to be a potential participants in this study
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
overall stability index | 3 months
  overall stability index was measured by using biodex balance system. by asking each participant to stand on biodex plateform trying to keep his balance while standing on one leg

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University For Science and Technology, Gamasa, Egypt